CLINICAL TRIAL: NCT00694928
Title: Vaginal Infection Study 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBC-303-603-622467
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis | interventions — clindamycin phosphate; butoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): clindamycin phosphate/butoconazole nitrate
  Interventions: Drug: clindamycin phosphate/butoconazole nitrate
- 2 (Active Comparator): butoconazole nitrate
  Interventions: Drug: butoconazole nitrate

INTERVENTIONS:
Drug: clindamycin phosphate/butoconazole nitrate — semi-solid, single dose
  Arms: 1
Drug: butoconazole nitrate — semi-solid, single dose
  Arms: 2

SUMMARY:
This study will evaluate the efficacy and safety of a vaginal product compared with that of another vaginal product in the treatment of vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of vaginal infection.
* Patients must be post-menopausal, surgically sterilized or using an acceptable form of birth control.

Exclusion Criteria:

* Patients must not have any other infections
* May not be pregnant or nursing
* May not be receiving any other antimicrobial therapies or any medications that would interfere with the outcome of the study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical symptom resolution | baseline, 7 to 10 days and 21 to 30 days

SECONDARY OUTCOMES:
Yeast Culture for Candida | baseline, 7 to 10 days and 21 to 30 days
  Negative Yeast Culture for Candida result=response, Positive Yeast Culture for Candida result=no response
Gram Stain Nugent Score | baseline, 7 to 10 days and 21 to 30 days
  Gram stain Nugent score of less than 4= resolution, Gram stain Nugent score of greater than 4= no resolution
Saline wet mount for clue cells | baseline, 7 to 10 days and 21 to 30 days
  Saline wet mount negative for clue cells=resolution, Saline wet mount positive for clue cells=no resolution

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Lumara Health, Inc.
Locations (73):
- United States (43):
  - Brookwood Ob-GYN, PC/Women's Medical Plaza, Birmingham, Alabama
  - Drug Research Analysis Corp, Montgomery, Alabama
  - Drug Research and Analysis Corp., Montgomery, Alabama
  - Ob/Gyn Associates, Jonesboro, Arkansas
  - The Woman's Clinic, PA, Little Rock, Arkansas
  - Peak Health Medical Group, Los Angeles, California
  - Women's Health Care at Frost Street, San Diego, California
  - Steven Freedman, MD, Inc., West Hills, California
  - Red Rocks OB/GYN, Lakewood, Colorado
  - SHE Medical Center, Hartford, Connecticut
  - Debra Hemsath, MD, Largo, Florida
  - International Research Associates, Miami, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - University Clinical Research, Pines, Florida
  - Total Women's Health and Wellness, Decatur, Georgia
  - Dekalb Gynecology Associates, Decatur, Georgia
  - New Millennium Ob/Gyn, Riverdale, Georgia
  - The Woman's Clinic, Boise, Idaho
  - The Iowa Clinic Department of Ob/Gyn, West Des Moines, Iowa
  - Steven Z. Lenowitz, MD, LLC, Bel Air, Maryland
  - Lawrence Ob/Gyn Associates, Lawrenceville, New Jersey
  - Women's Health Research Center, LLC, Lawrenceville, New Jersey
  - Triangle Ob/Gyn, Cary, North Carolina
  - Women's Wellness Center, Fayetteville, North Carolina
  - Meridian Clinical Research, LLC, Greensboro, North Carolina
  - Holzer Clinic, Gallipolis, Ohio
  - Family Practice Center of Wadsworth, Inc, Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Pacific Women's Center, LLC/Clinical Trials of America, Eugene, Oregon
  - Center for Women's Health of Lansdale, Lansdale, Pennsylvania
  - Creekside Women's Care, Charleston, South Carolina
  - The Family Healthcare Center, PA, Clinton, South Carolina
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - James T. Martin, Jr., MD, Ob/Gyn, North Charleston, South Carolina
  - Brown Clinical, PLLP, Watertown, South Dakota
  - Gynecology and Obstetrics, Memphis, Tennessee
  - Mid-South Ob/Gyn, Memphis, Tennessee
  - Kaner Medical Group, PA, Euless, Texas
  - Advanced Reserch Associates, McAllen, Texas
  - Willowbend Health & Wellness, Plano, Texas
  - Taylor/Wade Medical, Bountiful, Utah
  - Vermont Urogynecology Associates, PC, Williston, Vermont
  - Tidewater Clinical Research, Virginia Beach, Virginia
- India (10):
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - AJ Medical College and Hospital, Mangalore, Karnataka
  - Mayani Hosptial and Research Centre, Ajmer, Rajasthan
  - Sharda Hospital, Jaipur, Rajasthan
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Care Hospital, Hyderabad
  - Shri Krishna Hospital, Jaipur
  - Mediciti Institute of Medical Sciences, Ranga Reddy District
  - Krishna Institute of Medical Sciences, Secunderabad
  - King George Hospital, Visakhapatnam
- Russia (20):
  - Kurortniy Ward City Hospital #40, Sestroretsk, Sankt-Peterburg
  - Medical University Clinic, Kazan'
  - Clinical Dermatovenerologic Dispensary, Krasnodar
  - State Dermatovenerology Research Center of the Federal Agency for Provision of High Technology Medical Aid, Moscow
  - State Health Care Institution Moscow City Clinical Hospital #12, Moscow
  - Russian Medical Academy of Postgraduate Studies of Roszdrav, Moscow
  - State Healthcare Institution Moscow Clinical Hospital #68, Moscow
  - Novisibirsk Municipal Dermatovenerologic Dispensary #1, Novosibirsk
  - State Health Care Institution Orenburg Regional Clinical Hospital #2, Orenburg
  - Republican Dermatovenerologic Dispensary, MoH of Karelia Republic, Petrozavodsk
  - Maximillian City Hospital #28, Saint Petersburg
  - State Healthcare Institution Regional Dermatovenerologic Dispensary, Saint Petersburg
  - S.M. Kirov Military Medical Academy, MoD of the Russian Federation, Saint Petersburg
  - City Multifield Hospital, Saint Petersburg
  - Medical Research Institute, LLC, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - St. Petersburg I.P. Pavlov State Medical University of Roszdrav, Saint Petersburg
  - Railway Clinic Hospital of the Voronezh-,1 Railway Station, RJD JSC, Voronezh
  - Voronezh Regional Clinical Dermatovenerologic Dispensary, Voronezh
  - Yaroslavl Regional Maternity Hospital, Yaroslavl